CLINICAL TRIAL: NCT01430390
Title: A Phase I Trial Using In Vitro Expanded Allogeneic Epstein-Barr Virus Specific Cytotoxic T-Lymphocytes (EBV-CTLs) Genetically Targeted to the CD19 Antigen in B-cell Malignancies
Brief Title: In Vitro Expanded Allogeneic Epstein-Barr Virus Specific Cytotoxic T-Lymphocytes (EBV-CTLs) Genetically Targeted to the CD19 Antigen in B-cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-038
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphocytic Leukemia; Lymphoma
Keywords: In Vitro Expanded Allogeneic Epstein-Barr Virus Specific Cytotoxic; T-Lymphocytes (EBV-CTLs); CD19 specific T-cells; 11-038
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — Biological Products

STUDY DESIGN:
Intervention Model Description: This is a phase I trial designed to identify tolerable and clinically active doses of allogeneic Epstein - Barr virus specific cytotoxic T lymphocytes (EBV-CTLs) genetically modified to target the B-cell antigen CD19 when administered to patients with CD19+

ARMS (1):
- Biological/Genetically Modified T cells (Experimental): Utilizing our initial trial experience, it was amended to include three (3) expansion cohorts. Cohort 1: patients with CD19+ relapse/refractory (R/R) B cell malignancies occurring after allogeneic/autologous HSCT or solid organ transplant (SOT) infusion occurring following conditioning chemotherapy. Cohort 2:patients with CD10+ high risk B cell malignancies eligible for autologous HSCT followed by 19-28z CRA EBV-CTLs (auto-HSCT preparative regimen serves as conditioning chemotherapy. Cohort 3: patients with CD19+ high risk B cell malignancies eligible for allogeneic HSCT followed by consolidative 19-28z CAR EBV-CTLs (allo-HSCT preparative regimen serves as conditioning chemotherapy) Each expansion cohort has a target accrual of 6 patients treated with fixed CAR EBV-CTL dose (3x106 EBV-CTLs/kg) which has been demonstrated to be the ideal manufacturing dose.
  Interventions: Biological: Biological/Genetically Modified T cells; Drug: Cyclophosphamide-based chemotherapy

INTERVENTIONS:
Biological: Biological/Genetically Modified T cells — Following completion of the chemotherapy, genetically modified T cells will be given intravenously at one of 3 dose levels. After the infusion patients will be monitored clinically and with serial blood and marrow evaluations to assess toxicity, therapeutic effects, and the in-vivo survival of the genetically modified T-cells. A fixed CAR EBV-CTL dose (3x106 EBV-CTLs/kg) which has been demonstrated to be the ideal manufacturing dose allowing for multiple infusions and potential for multiple patient treatments per cell line generated will be used for all patients on this trial. Cohorts will be determined separately but cohort 3 will not begin to accrue until cohort 2 has treated three (3) patients without a DLT. Each patient is eligible for up to three (3) infusions.
Drug: Cyclophosphamide-based chemotherapy — Cyclophosphamide-based chemotherapy regimen will be the preferred conditioning chemotherapy prior to CAR T cell infusion for patients with CD19+ malignancy in cohort 1. Recommended chemotherapy regimen consists of single agent Cyclophosphamide at a dose of 3000 mg/m2/dose IV over 1 hour or 1500mg/m2/dose x 2 doses given daily over 1 hour given for 2 days (patients may received reduced dose of cyclophosphamide based on the clinical status of the patient at discretion of the treating physician and with written approval by the MSKCC PI of this study). Alternative cyclophosphamide or non-cyclophosphamide-based regimens based on the clinical status of the patient, disease burden, and likely-hood of response may be used at the discretion of the treating physician with written approval by MSKCC PI of the study. Conditioning chemotherapy will not be given prior to infusions # 2 and #3.

SUMMARY:
The purpose of this study is to test the safety of giving the patient special cells from a donor called "Modified T-cells". The goal is to assess the toxicities of T-cells for patients with relapsed B cell leukemia or lymphoma after a blood SCT organ SCT or for patients who are at high risk for relapse of their B cell leukemia or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* History of CD19+ relapse/refractory (R/R) B cell malignancies occurring after allogeneic/autologous HSCT or solid organ transplant (SOT. (cohort 1)
* Relapse on this protocol is detection of CD19+ malignancies in bone marrow morphology ≥ 5% any extramedullary lesion (radiographic), or detection of any disease level by cytogenetics, molecular, and/or flow cytometry.
* History of relapsed or refractory CD19+ malignancies (e.g. Non Hodgkin Lymphoma) or considered high risk for relapse and and require autologous or allogeneic hematopoietic stem cell transplant (HSCT). Evidence of disease not required. (cohort 2 and 3)
* No age restriction for patients
* KPS or Lansky score > or = to 50
* Renal function (measured prior to conditioning chemotherapy)
* Creatinine ≤ 2.0mg/dL for patients over 18 years of ≤ 2.5 x institutional ULN for age.
* Hepatic function (measured prior to conditioning chemotherapy):
* AST ≤ 5 x the institutional ULN Elevation secondary to leukemic involvement is not an exclusion criterion. Leukemic involvement will be determined by the presence of progressive relapse defined by escalating bone marrow or peripheral blood leukemia blasts within the previous month and the absence of initiation of know hepatotoxic medication (e.g. azoles).
* Total bilirubin ≤ 2.5 x the institutional ULN
* Adequate cardiac function (e.g. LVEF ≥ 40%) as assessed by ECHO or MUGA or other similar cardia imaging performed within 1 month of treatment.
* Pulmonary function (measured prior to treatment):
* Oxygen saturation ≥ 90% on room air

Donor Eligibility:

* The patient's HSCT donor, or if HSCT donor is not available a third party donor, must consent to a leukapheresis or whole blood donation(s) obtained at one or more phlebotomies which, in aggregate, will total approximately 250 ml for adults and no more than 5ml/kg per draw from pediatric donors.
* Related donors <18 years of age requiring placement of a leukapheresis catheter will donate peripheral blood collected by phlebotomy (including a unit of blood if weight permits) and shall not undergo catheter placement for leukapheresis as this is considered above minimal risk to the donor.
* There is no upper age limit for a donors. However, the minimum age for a related donor is 7 years as this is the youngest age a person can be considered capable of giving assent to participate in a research study.
* Evidence of prior sensitization to EBV by EBV serology testing (seropositive)
* Donor's high resolution HLA typing must be available for review
* CBC within one week of donation. Results of tests must be within a range that would not preclude donating blood or undergoing leukapheresis.
* Serologic testing for transmissible diseases will be performed as per institutional guidelines adopted from extant NMDP and FACT guidelines. Donors should be considered eligible to donate leukapheresis or blood based on these guidelines (i.e. blood donation guidelines)

Exclusion Criteria:

* Patients with active HIV, hepatitis B or hepatitis C infection.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation.
* Females who are pregnant.
* Patients will be excluded if they have isolated extra-medullary relapse of ALL.
* Patients with active (grade 2-4) acute graft versus host disease (GVHD), chronic GVHD or an overt autoimmune disease (e.g. hemolytic anemia) requiring glucocorticosteroid treatment (>0.5 mg/kg/day prednisone or its equivalent) as treatment
* Active central nervous system (CNS) leukemia, as defined by unequivocal morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF) or symptomatic CNS leukemia (i.e. cranial nerve palsies or other significant neurologic dysfunction) within 28 days of treatment. Prophylactic intrathecal medication is not a reason for exclusion.
* Adult patients (≥18 years old) with the following cardiac conditions will be excluded:
* New York Heart Association (NYHA) stage III or IV congestive heart failure
* Myocardial infarction ≤ 6months prior to enrollment
* History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration.
* History of severe non-ischemic cardiomyopathy with EF ≤20%
* Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the treating investigator would pose an unacceptable risk to the subject.
* Prior irreversible neurologic toxicity to previous immunotherapy
* Preceding and/or ongoing organ dysfunction or other co-morbidity including but not limited to uncontrolled infection that would impair the patient's ability to endure known side effects of cytokine release syndrome or neurological toxicity
* Recent prior therapy: Systematic chemotherapy less than 2 weeks prior to infusion.
* Recent prior therapy: Systematic chemotherapy less than 2 weeks prior to infusion. Exceptions:

  * There is no time restriction in regard to prior intrathecal chemotherapy provided tere is complete recovery from any acute toxic effects of such.
  * Subjects receiving hydroxyurea or oral maintenance chemotherapy may be enrolled provided there has been no increase in dose for at least 2 weeks prior to starting apheresis or treatment
  * Subjects receiving steroid therapy at physiological replacement doses only are allowed provided there has been no increase in dose for at least 2 weeks prior to subject starting apheresis or treatment.
  * Subjects must have recovered from the acute side effects of their prior therapy, such that eligibility criteria are met. Cytopenias deemed to be disease-related and not therapy-related are exempt from this exclusion.
* Rapidly progressive disease that in the estimation of the treating physician would compromise ability to complete study therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety/persistence of (including GVHD) of allogeneic EBV specific CTL modified to express artificial T cell receptors targeting CD19 molecule given for persistence or relapse of B-Cell ALL post allogeneic HSCT. | 3 years

SECONDARY OUTCOMES:
To assess the effects of the adoptively transferred CD19 specific T-cells on the progression of leukemia. | 3 years
To quantitate the number of chimeric antigen receptor (CAR) positive T-cells and donor EBV-CTL in the blood at defined intervals post infusion in order to determine their survival and proliferation in the host. | 3 years
To assess long-term status of treated patients | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Curran, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Shahid S, Prockop SE, Flynn GC, Mauguen A, White CO, Bieler J, McAvoy D, Hosszu K, Cancio MI, Jakubowski AA, Scaradavou A, Boelens JJ, Sauter CS, Perales MA, Giralt SA, Taylor C, Chaudhari J, Wang X, Riviere I, Sadelain M, Brentjens RJ, Kernan NA, O'Reilly RJ, Curran KJ. Allogeneic off-the-shelf CAR T-cell therapy for relapsed or refractory B-cell malignancies. Blood Adv. 2025 Apr 8;9(7):1644-1657. doi: 10.1182/bloodadvances.2024015157. PMID 39908482
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm